CLINICAL TRIAL: NCT05211076
Title: The Effect of Music Practice and Marmet Technique on Lactation and Maternal Anxiety in Mothers With Premature Babies: A Randomized Controlled Study
Brief Title: The Effect of Music Practice and Marmet Technique on Lactation and Maternal Anxiety in Mothers With Premature Babies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Resmiye KAYA ODABAŞ (Other)
Collaborators: Goztepe Training and Research Hospital (Other); Uşak University (Other)
Responsible Party: Sponsor-Investigator, Resmiye KAYA ODABAŞ, Principal Investigator, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: resmiye-0001
Record Dates: First submitted 2022-01-12; First posted 2022-01-27 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Lactation
Keywords: lactation; marmet technique; music therapy; maternal anxiety; breast milk; nonpharmacological method
MeSH Terms: conditions — Breast Feeding | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Group (Experimental): In the selection of the music to be played,Rast,Uşşak,Kürdi,Muhayyer modes were chosen by taking expert opinion.Before starting the music application,the selected music will be sent to the mothers in this group by the researcher over the internet to the mother's phone and it will be ensured that the mother listens to the music transmitting the sound from her own phone in each session.
  * Music practice will take place in mothers' rooms or in the NICU.
  * The room will be quiet and your mother will be alone.
  * To make the mother listen to music;The mother will be asked to sit on the bed/seat in a comfortable position.
  * At the same time,the mother will be asked to close her eyes and be relaxed.
  * Later, music will be turned on from the mother's phone, allowing the mother to listen to music for 30 minutes
  * While the mother listening to the music,at the 16th minute of the music,researcher will manually express each breast separately for at least 15 minutes until no milk comes out
  Interventions: Other: Music Group
- Marmet Technique Group (Experimental): Marmet Technique is one of the non-pharmacological methods used to increase milk production.The Marmet Technique is a combined method that includes breast massage and manual milking.The Marmet Technique will be performed in the mothers' rooms or in the Breastfeeding Room of the Neonatal Intensive Care Unit. It will be ensured that the mother is comfortable by paying attention to her privacy. Mothers will be manually milked into the hopper in their own milking set. In addition, the reservoir will be used after washing with hot water. This technique consists of two stages, these stages are emptying the milk ducts and stimulating the milk stroke reflex (massage).
  Interventions: Other: Marmet Technique Group
- control group (Experimental): On the other hand, no application will be made to the control group, and the milking process will be carried out manually by the researcher for at least 15 minutes until the milk does not come.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Music Group — The Introductory Information Form will be filled in by researcher using face-to-face interview technique.It will be ensured that the mother fills the State Anxiety Scale with her own statement.On the 1st day of the post-op,mothers will be able to listen to Classical Turkish Music works in the forms of Saz Semaisi,Peşrev,Medhal in Rast,Uşşak,Kürdi,Muhayyer makams for 30 minutes via their phone at 11:00am.
  While the mother continues to listen to the music,at the 16th minute,the researcher will manually milk the mother for at least 15 minutes until milk comes out.At the end of the milking process,the milk accumulated in the container will be measured by the researcher with injector,recorded in the Breast Milk Follow-up Form.At the end of the music session,it will be ensured that the mother fills in the State Anxiety Scale with her own statement.
  The same procedure will be applied to the mother atb05:00pm.This process will be carried out 8 times in total,at 11:00am and 05:00pm for 4days.
  Arms: Music Group
Other: Marmet Technique Group — Consent will be obtained from those who agree to participate in the study. The Introductory Information Form will be filled by the researcher using face-to-face interview technique.
  It will be ensured that the mother fills the State Anxiety Scale with her own statement.
  The Marmet Technique will be applied to the mothers at 11:00am for 20-30 minutes by the researcher.
  At the end of the milking process performed in accordance with the technique, the milk accumulated in the container will be measured with an injector and recorded in the Breast Milk Follow-up Form.
  Then, it will be ensured that the mother fills in the State Anxiety Scale with her own statement.
  At 05:00pm, the same procedure will be applied to the mother. At the end of the 4th day, the satisfaction of the mother will be evaluated on the Mother Satisfaction Evaluation Scale.This process will be carried out 8 times in total,at 11:00am and 05:00pm for 4days.
  Arms: Marmet Technique Group
Other: Control group — The Introductory Information Form will be filled by the researcher using face-to-face interview technique.It will be ensured that the mother fills the State Anxiety Scale with her own statement.The mothers will milk the mother manually by the researcher at 11:00am for at least 15 minutes until the milk does not come.
  At the end of the milking process, the milk accumulated in the container will be measured with an injector and recorded in the Breast Milk Follow-up Form in ml.
  Then, it will be ensured that the mother fills in the State Anxiety Scale with her own statement. At 05:00pm, the same procedure will be applied to the mother.
  At the end of the 4th day, the satisfaction of the mother will be evaluated on the Mother Satisfaction Evaluation Scale.This process will be carried out 8 times in total,at 11:00am and 05:00pm for 4days.
  Arms: control group

SUMMARY:
This study was planned as a randomized controlled study to examine the effect of music practice and Marmet Technique on lactation and maternal anxiety in mothers with premature babies in the neonatal intensive care unit.The research will be carried out with 32+0 and 36+6 weeks old preterms hospitalized in the Suleyman Yalçin City Hospital NICU.It will be held between January and December 2022 with mothers of premature babies born by cesarean section between weeks of gestation.The research will be carried out with three groups as music,Marmet Technique and control group.The sample number was calculated using the G*Power program and the music group:22,the Marmet Technique:22,and the control group: 22 (n=66).It is planned to collect the data with the Introductory Information Form, the Breast Milk Follow-up Form, the State Anxiety Scale and the Maternal Satisfaction Evaluation Scale.Post-op with mothers on day 8-12. Information about the research will be given by meeting between hours and written and verbal consent will be taken.Randomization will be applied to the mothers who accepted the study.During the study,all mothers will be informed that music and Marmet Technique will be performed at 11:00 and 17:00, 2 sessions a day for 4 days,starting from the post-op day 1,and then the milking process will be performed,and the mothers will be provided to come to the breastfeeding room at the specified times.The State Anxiety Scale will be filled in by the mother,and then the music will be played for 15 minutes.In the 16th minute,milking will be performed manually by the researcher and the milking process will take at least 15 minutes.After the milking process,the mother will fill the State Anxiety Scale again.In the Marmet Technique group,the State Anxiety Scale will be filled first by the mother,and then massage and milking will be performed for 20-30 minutes in accordance with the protocol of the technique.After the milking process,the mother will fill in the State Anxiety Scale again.No application will be made to the control group. Breast milk will be provided manually by the researcher for at least 15 minutes.The data of the research will be evaluated using the SPSS program.In the evaluation of the data;descriptive statistics will be done with One Way Analysis of Variance Kruskal Wallis H Test.In order to determine the difference in milk amounts between groups,repeated measure covariance analysis will be applied.

DETAILED DESCRIPTION:
Primary aim: The primary purpose of the study is to examine the effects of music practice and Marmet Technique on lactation and maternal anxiety in mothers with premature babies.

Secondary aim: The secondary aim of the research is to contribute to the literature on music practice and Marmet Technique.

Hypotheses:

H0: There is no difference in the amount of breast milk between the music, Marmet Technique and control groups in mothers with premature babies in the neonatal intensive care unit.

H1: There is a difference in the amount of breast milk between the music, Marmet Technique and control groups in mothers with premature babies in the neonatal intensive care unit.

H0: There is no difference in maternal anxiety between music, Marmet Technique and control groups in mothers with premature babies in the neonatal intensive care unit.

H1: There is a difference in maternal anxiety between music, Marmet Technique and control groups in mothers with premature babies in the neonatal intensive care unit.

This study was designed as a randomized controlled experimental study. The study was conducted at the Suleyman Yalçin City Hospital from January to December 2022.

The universe of the research is Göztepe Prof. Dr. 32+0- and 36+6 patients hospitalized in the Newborn Intensive Care Unit of Suleyman Yalçin City Hospital. Mothers of premature babies born before the week of gestation will form. The research will be carried out with three groups as music, Marmet Technique and control group. Sample size, according to to examine the effect of listening to music on postpartum depression and lactation. The sample size of the study was calculated using the G*Power 3.1.9.2 program and the mean, standard deviation and sample size values of the breast milk variable included in the related article were taken into account in calculating the effect size. In the music group, the mean and standard deviation values of the breast milk variable were 60.50±25.30 and n=30. In the control group, the mean and standard deviation values of the breast milk variable were 31.30±22.60 and n=30. Using the mean, standard deviation and sample number values of the related article, the mean standard deviation value was found to be 23.98, and as a result, the effect size was calculated as 0.60. The minimum number of individuals to be included in the sample of this study was calculated by taking G*Power 3.1.9.2 and f: 0.60, α= 0.05, 1-β: 0.95, and the sample size was determined as at least 45 mother (15 mother for each group). In order to increase the analysis power, the number of samples was increased and n=22 was taken for each group (music group: 22, marmet technique group: 22 and control group: 22). In which group the mothers included in the study will be, will be determined from the website of the random number generation program "Research Lists", and they will be divided into three groups.

Randomization: The group that the mothers will be in is determined from the random number generation website called "Random Lists". The mothers were divided into three groups as the music group, the Marmet Technique group and the control group. Thus, each mother's number will be determined and recorded.

Research data, Descriptive Information Research data, Descriptive Information Form, Breast Milk Follow-up Form, State Anxiety Scale and Maternal Satisfaction Evaluation Scale will be collected.

Introductory Information Form: This form was prepared by the researchers in line with the literature.There are 26 questions in the form, including socio-demographic (5), obstetric characteristics (5), general health information (7), characteristics related to breast milk and breastfeeding (4), and newborn characteristics (5).

Breast Milk Follow-up Form: For each day, in this form prepared by the researchers; Information about the time elapsed since the last milking, the duration of milking, the amount of milk expressed, the daily sleep duration of the mother and the amount of fluid consumed by the mother are included.

State Anxiety Inventory: The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely. A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered as the lowest level of anxiety and 80 as the highest level of anxiety.

Maternal Satisfaction Evaluation Scale: In this scale, which was prepared by the researchers, it was aimed to evaluate the satisfaction of mothers regarding the practices performed by scoring between 0-10. It is expressed as 0: "Not at all satisfied" and 10: "Very satisfied, satisfied".

Preliminary work will be done with five mothers before starting the study in order to assess whether the questions have been understood. As a result of the evaluation, it will be evaluated whether there is a need for editing in the data forms and adjustments will be made. Those included in the pilot application will not be included in the sample group.

Data Collection In order to carry out the study, after obtaining the permission of the ethics committee and the institution, the mothers who performed cesarean section will be met on the 0th post-op day by going to the institution. The mothers who meet the research criteria will be informed about the purpose, content and methods of the research and those who want to participate in the study will be determined. Then, in which group the mothers will be, they will be divided into three groups as music, Marmet Technique and control group through the random number generation program "Random Lists". Thus, each mother's number will be determined and recorded. Verbal and written consent will be obtained from those who accept the study. Since the mothers had pain on the post-op day 0, it is planned to start the study at 11:00 on the post-op 1st day.

In the study, the data will be filled in by the researcher working as a midwife in the Neonatal Intensive Care Unit in the same hospital, by face-to-face interview technique in the Breastfeeding Room of the Neonatal Intensive Care Unit. During the study, all mothers will be informed that music practice and Marmet Technique will be performed at 11:00 and 17:00, 2 sessions a day (8 sessions in total) for 4 days, and then the milking process will be performed, and it will be ensured that the mothers come to the breastfeeding room at the specified times. Depending on the mother's condition, the application and milking process will be carried out in the patient's room during the hospitalization, or in the Breastfeeding Room of the Neonatal Intensive Care Unit for those who can come to the breastfeeding room.

First of all, the State Anxiety Scale for the music group will be filled by the mother and then the music will be played for 15 minutes. While the music continues, milking will be performed manually by the researcher at the 16th minute and the milking process will take at least 15 minutes (music listening time will take 30 minutes in total). After the milking process, it will be ensured that the mother fills in the State Anxiety Scale again. In the Marmet technique group, the State Anxiety Scale will be filled by the mother first, and then massage and milking will be performed for 20-30 minutes in accordance with the protocol of the technique. After the milking process, the mother will have to fill in the State Anxiety Scale again. On the other hand, no application will be made to the control group, and milking will be performed manually by the researcher for at least 15 minutes until the milk does not come.

It will be ensured that the mother completes the State Anxiety Scale before and after the milking process. Applications and milking process,

1. st day 2 times,
2. st day 2 times,
3. st day 2 times,
4. st day 2 times, The milking process will be carried out by performing music and Marmet Technique separately for each group, 8 times in total. No application will be made to the control group, and only the milking process and the filling of the forms will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* In the 18-35 age range,
* Primiparous and multiparous,
* Birth by cesarean section between 32+0 and 36+6 gestational weeks,
* The baby is hospitalized in the Neonatal Intensive Care Unit,
* Babies who cannot be breastfed, but fed and tolerated by gavage,
* Willing to feed their baby with breast milk,
* Able to speak and understand Turkish,
* The mothers who agreed to participate in the study

Exclusion Criteria:

* Having advanced congenital anomaly in her baby,
* Babies with contraindications for breastfeeding (galactosemia, congenital anomalies, etc.),
* Having any health problems (tuberculosis, HIV, cancer, etc.),
* Having multiple pregnancies,
* Body mass index over 30,
* Those who became pregnant with infertility treatment,
* Using drugs to increase breast milk, vitamins and additional supplements,
* Having postpartum complications (bleeding, embolism, etc.),
* The baby and/or own Covid-19 positive,
* Mothers who smoke or drink alcohol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-01-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
amount of breast milk | On the 1st postoperative day, at 11:00 am.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 1st postoperative day, at 05:00 pm.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 2st postoperative day, at 11:00 am.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 2st postoperative day, at 05:00 pm.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 3st postoperative day, at 11:00 am.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 3st postoperative day, at 05:00 pm.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 4st postoperative day, at 11:00 am.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
amount of breast milk | On the 4st postoperative day, at 05:00 pm.
  The amount of breast milk will be expressed manually for at least 15 minutes until no milk comes out.
  At the end of the milking process, the amount of milk accumulated in the container will be measured by the researcher with an injector and recorded in the Breast Milk Follow-up Form in milliliters and delivered to the newborn midwife/nurse.
State Anxiety Scale | Pre-intervention at 11:00 am on the postoperative 1st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 11:00 am on the postoperative 1st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 05:00 pm on the postoperative 1st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 05:00 pm on the postoperative 1st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 11:00 am on the postoperative 2st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 11:00 am on the postoperative 2st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 05:00 pm on the postoperative 2st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 05:00 pm on the postoperative 2st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 11:00 am on the postoperative 3st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 11:00 am on the postoperative 3st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 05:00 pm on the postoperative 3st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 05:00 pm on the postoperative 3st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 11:00 am on the postoperative 4st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 11:00 am on the postoperative 4st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Pre-intervention at 05:00 pm on the postoperative 4st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.
State Anxiety Scale | Post-intervention at 05:00 pm on the postoperative 4st day.
  The scale, which consists of 20 questions in total, determines how the individual feels at the moment. Behaviors and emotions expressed in the items of the scale are marked as (1) none, (2) a little, (3) a lot, and (4) completely (Öner & Le Compte, 1983). A total score is obtained and an evaluation is made over a minimum of 20 and a maximum of 80 points. In addition, there are reversed and direct/straight statements in the scale, and a 4 point answer in direct statements indicates high anxiety. In reversed statements, answers with 1 point indicate a high level of anxiety. Items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20 are reversed statements. In these items, 1 point is given 4 points, 2 points 3 points, 3 points 2 points, 4 points 1 point. In the scoring of the scale, the level of anxiety increases as the scores increase, and 20 is considered the lowest level of anxiety and 80 the highest level of anxiety.

SECONDARY OUTCOMES:
Maternal Satisfaction Rating Scale | Post-intervention at 05:00 pm on the postoperative 4st day.
  In this scale prepared by the researchers, it was aimed to evaluate the satisfaction of the mothers regarding the practices performed by scoring between 0-10. 0: "Not at all satisfied" and 10: "Very satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Hüsnü Fahri OVALI, Prof. Dr., Principal Investigator — Goztepe Training and Research Hospital; Ayla ERGİN, Ass.Prof., Study Director — Kocaeli University; Şeyma ÇATALGÖL, Instructor, Study Chair — Uşak University; Ebru Aktaş, Midwifery, Study Chair — Goztepe Training and Research Hospital
Locations (1):
- Prof. Dr. Süleyman Yalçın City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No